CLINICAL TRIAL: NCT04813679
Title: Bed-side Ultrasound in the Evaluation of Gastro-intestinal Tract and Neutropenic Enterocolitis (NEC) in Neutropenic Patients.
Brief Title: Bed-side Ultrasound in Neutropenic Enterocolitis
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Edoardo Benedetti, Medical director, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: NEC_3636
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Neutropenic Enterocolitis
Keywords: NEC, bed side ultrasound, diagnosis, treatment
MeSH Terms: conditions — Enterocolitis, Neutropenic; Enterocolitis, Necrotizing; Disease | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neutropenic Enterocolite patients assessed with bed side ultrasound sonography: From March 2007 through the entire study period all patients admitted eighter in our chemotherapy-ward or BMT-ward to receive intensive chemotherapy (chemo) for any hematological malignancies, or chemotherapy (CHT) for both auto transplant (ASTC) and allogeneic transplant (AlloTx), were prospectively enrolled in the study. When the patient received more than one chemo cycle, each ward access was considered a new observational period.
  Patients who received CHT and experienced CHT-induced neutropenia (CHTNP) were enrolled in the study. We defined "one observational period" each admission on the ward to receive CHT, in which CHT and length of stay could vary from the previous admission. One observational period ended with the discharge of the pts form the ward. If a pts experienced a new chemo related NECe during another admission, it was considered as e new NECe.
  Interventions: Diagnostic Test: Bed side Ultrasound Sonography
- Neutropenic Enterocolite negative patients assessed with bed side ultrasound sonography: NEC negative patients received bed-side ultrasound sonography after three days of neutropenia.
  Interventions: Diagnostic Test: Bed side Ultrasound Sonography

INTERVENTIONS:
Diagnostic Test: Bed side Ultrasound Sonography — Bed side Ultrasound in Neutropenic patients within 12 h from onset of any symptom such as fever and/or abdominal pain and/or diarreha
  Other Names: imaging

SUMMARY:
Neutropenic enterocolitis (NEC) is a life-threatening complication of leukemic and solid tumors patients (pts) treated with chemotherapy (CHT) with high mortality rate up to 50-100%. Perforation occurs in 5%-10% of cases. Early diagnosis is crucial to start conservative medical management (CMM), which appears the optimal strategy for most cases.

NEC should be always suspected in Neutropenic pts with abdominal pain, fever and diarrhea.

Ultrasound (US) can be used to evaluate bowel-wall thickening (BWT). The objective of this study is to evaluate prospectively if US can detect early signs of NEC and guide a prompt treatment (CMM or surgical) and thus reduce mortality.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted in Hematology Ward University of Pisa (Italy) to receive chemotherapy who experienced neutropenia related to chemotherapy

Exclusion Criteria:

Patients admitted in Hematology Ward University of Pisa (Italy) who did not receive chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in Hematology Ward University of Pisa (Italy) from March 2007 to January 2018 to receive chemotherapy who experienced neutropenia related to chemotherapy, were prospectively enrolled
Sampling Method: Non-Probability Sample
Enrollment: 1740 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
to verify the hypothesis that US could detect early signs of NEC, guide a prompt treatment eventually reducing mortality | from March 2007 to January 2018
  Bed side Ultrasound sonography assessment of bowel in neutropenic patients with fever and/or abdominal pain and/or diarrhea
to correlate patient's symptoms with outcome | from March 2007 to January 2018
  Statistical correlation of symptoms with outcome
to verify if bowel wall thickening (BWT) is pathognomonic of neutropenic enterocolitis | from March 2007 to January 2018
  Comparison of bowel wall thickness in patients with diagnosis of neutropenic enterocolitis and in the control group (NEC negative group)
to find which symptom or symptoms have a higher relative risk (RR) for NEC diagnosis | from March 2007 to January 2018
  Statistical analysis of symptoms in the NEC group at diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Unit, Santa Chiara Hospital University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benedetti E, Bruno B, McDonald GB, Paolicchi A, Caracciolo F, Papineschi F, Pelosini M, Campani D, Galimberti S, Petrini M. Prospective qualitative and quantitative non-invasive evaluation of intestinal acute GVHD by contrast-enhanced ultrasound sonography. Bone Marrow Transplant. 2013 Nov;48(11):1421-8. doi: 10.1038/bmt.2013.65. Epub 2013 May 13. PMID 23665821
- [Background] Benedetti E, Tavarozzi R, Morganti R, Bruno B, Bramanti E, Barate C, Balducci S, Iovino L, Ricci F, Ricchiuto V, Buda G, Galimberti S. Organ Stiffness in the Work-Up of Myelofibrosis and Philadelphia-Negative Chronic Myeloproliferative Neoplasms. J Clin Med. 2020 Jul 8;9(7):2149. doi: 10.3390/jcm9072149. PMID 32650390
- [Background] Benedetti E, Barate C, Bruno B, Bramanti E, Ghia P, Scarfo L, Morganti R, Ricchiuto V, Galimberti S. Response assessment to venetoclax in relapsed/refractory chronic lymphocytic leukemia by ultrasonography. Leuk Res. 2021 Jan;100:106488. doi: 10.1016/j.leukres.2020.106488. Epub 2020 Nov 30. No abstract available. PMID 33316660
- [Background] Benedetti E, Proietti A, Miccoli P, Basolo F, Ciancia E, Erba PA, Galimberti S, Orsitto E, Petrini M. Contrast-enhanced ultrasonography in nodular splenomegaly associated with type B Niemann-Pick disease: an atypical hemangioma enhancement pattern. J Ultrasound. 2009 Sep;12(3):85-92. doi: 10.1016/j.jus.2009.06.001. Epub 2009 Jul 9. PMID 23396497
- [Background] Benedetti E, Lippolis PV, Caracciolo F, Galimberti S, Papineschi F, Pelosini M, Focosi D, Stella SM, Neri E, Seccia M, Petrini M. Ultrasound findings guided a successful hemicolectomy in a leukemic patient with neutropenic enterocolitis. J Ultrasound. 2008 Sep;11(3):97-101. doi: 10.1016/j.jus.2008.05.001. Epub 2008 Jul 3. PMID 23396752
- [Background] Di Franco G, Tagliaferri E, Pieroni E, Benedetti E, Guadagni S, Palmeri M, Furbetta N, Campani D, Di Candio G, Petrini M, Mosca F, Morelli L. Multiple small bowel perforations due to invasive aspergillosis in a patient with acute myeloid leukemia: case report and a systematic review of the literature. Infection. 2018 Jun;46(3):317-324. doi: 10.1007/s15010-018-1115-7. Epub 2018 Jan 22. PMID 29357049